CLINICAL TRIAL: NCT01997463
Title: The Cost Effectiveness of School-Based Supervised Asthma Therapy
Brief Title: Supervised Asthma Medication in Schools (SAMS)
Acronym: SAMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200000709; 1R18HL110858 (NIH)
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Results first posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Childhood Asthma
MeSH Terms: interventions — Schools; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular Therapy (No Intervention): Regular Asthma Therapy
- Supervised Therapy (Experimental): Supervised asthma therapy in schools
  Interventions: Drug: Supervised asthma therapy in schools

INTERVENTIONS:
Drug: Supervised asthma therapy in schools — Therapy observed daily in school. Asthma education by American Lung Association
  Other Names: Inhaled Corticosteroid; Ventolin
  Arms: Supervised Therapy

SUMMARY:
The investigators hypothesize that school-based, direct supervision of daily controller therapy will result in more effective asthma control, as assessed by the Asthma Control Questionnaire than usual care. Additionally, as the result of enhanced asthma control and resulting decrease in health care utilization, school-based, direct supervision of daily controller therapy will result in lower cost per quality-adjusted life year (QALY) gained than usual care.

DETAILED DESCRIPTION:
This research is being done to test if children with asthma will have fewer asthma symptoms if they are monitored at school to make sure they take their inhaled steroid medication (ICS) every day and take the medication the right way. All of the children with asthma in the school will be asked to participate. In the first year in one-half of the schools, children and school staff will participate in a standardized asthma education program presented by the American Lung Association (ALA). Children will have daily monitoring of their inhaled asthma medication. The other half of schools will continue with the usual treatment of children with asthma. In the second year of the study, all schools and children will have the asthma education program and monitoring. Parents will be queried quarterly for information about their child's asthma.

ELIGIBILITY:
Inclusion Criteria:

* A child with asthma attending a Tucson Unified School District elementary school selected for the study.

Exclusion Criteria:

* No asthma.
* Not attending a Tucson Unified School District elementary school selected for the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 442 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn B Gerald, Ph.D., MSPH, Principal Investigator — University of Arizona, Mel and Enid Zuckerman College of Public Health
Locations (1):
- The University of Arizona and the Tucson Unified School District, Tucson, Arizona, United States

REFERENCES:
- [Derived] Gerald JK, Fisher JM, Brown MA, Clemens CJ, Moore MA, Carvajal SC, Bryson D, Stefan N, Billheimer D, Gerald LB. School-supervised use of a once-daily inhaled corticosteroid regimen: A cluster randomized trial. J Allergy Clin Immunol. 2019 Feb;143(2):755-764. doi: 10.1016/j.jaci.2018.06.048. Epub 2018 Aug 14. PMID 30118728

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regular Therapy | Supervised Therapy
Started | 192 | 250
Completed | 107 | 147
Not Completed | 85 | 103

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regular Therapy | Supervised Therapy | Total
Number analyzed (Participants) | 192 | 250 | 442
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 192 | 250 | 442
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 88 | 160
  Male | 120 | 162 | 282
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 128 | 168 | 296
  Not Hispanic or Latino | 48 | 57 | 105
  Unknown or Not Reported | 16 | 25 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 32 | 44
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  Black or African American | 17 | 24 | 41
  White | 78 | 92 | 170
  More than one race | 62 | 66 | 128
  Unknown or Not Reported | 19 | 34 | 53

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be the Score on the Juniper Asthma Control Questionnaire (ACQ)
Description: An ACQ score of > 1.5 means asthma is not well controlled. An ACQ score of <= 1.5 means asthma is well controlled.
  Missing ACQ score = number of participants not administered an ACQ
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Regular Therapy | Supervised Therapy
Number analyzed (Participants) | 192 | 250
Participants
  Visit 1: ACQ score >1.5 (not well controlled) | 54 | 70
  Visit 1: ACQ score <=1.5(well controlled) | 74 | 95
  Visit 1: missing ACQ score | 64 | 85
  Visit 2: ACQ score >1.5 (not well controlled) | 56 | 73
  Visit 2: ACQ score <=1.5(well controlled) | 75 | 99
  Visit 2: missing ACQ score | 61 | 78
  Visit 3: ACQ score >1.5 (not well controlled) | 55 | 65
  Visit 3: ACQ score <=1.5(well controlled) | 75 | 116
  Visit 3: missing ACQ score | 62 | 69
  Visit 4: ACQ score >1.5 (not well controlled) | 60 | 65
  Visit 4: ACQ score <=1.5(well controlled) | 77 | 123
  Visit 4: missing ACQ score | 55 | 62

ADVERSE EVENTS:
Arm/Group | Regular Therapy | Supervised Therapy
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/250
Other Adverse Events (participants affected / at risk) | 0/192 | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No